CLINICAL TRIAL: NCT04283903
Title: Metabolomic and Proteomic Fingerprinting in Peri-implant Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: Metabol_Proteom_Implants
Record Dates: First submitted 2020-02-17; First posted 2020-02-25 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-12

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PICF — PICF collection from 4 sites

SUMMARY:
Due to the limited efficacy of its treatment modalities, there is a stringent need to improve the prevention and early diagnosis of peri-implantitis. In fact, to date clinical and radiographic tools are not able to discern which patients are going to develop peri-implantitis and, among the ones already with peri-implantitis, which ones are currently loosing bone and which ones are going to progress.

This project aims to analyze for the first time the whole large scale proteome and metabolome of peri-implant crevicular fluid (PICF) with an integrated approach from implants with peri-implant diseases.

Twenty-five patients with at least one implant with peri-implant mucositis and one implant with peri-implantitis will be selected. For each of the selected participants, the PICF from an implant with peri-implant mucositis and from an implant with peri-implantitis will be sampled two different times before treatment. One year after the corresponding treatment is provided, the PICF of the treated implants with peri-implantitis will be sampled again.

Both proteomic and metabolomic profiling of the samples will be carried out. The most important strength of this project will be the ability to evaluate together the whole proteome and the whole metabolome and to integrate them in the same framework.

ELIGIBILITY:
Inclusion Criteria:

* At least one implant with peri-implant mucositis and one with peri-implantitis

Exclusion Criteria:

* Previously treated implants to be included

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: According to a study with a similar design on periodontitis (Barnes et al. 2009), twenty-five patients with at least one implant with peri-implantitis and one implant with peri-implant mucositis (Berglundh et al. 2018) will be selected in Complutense University of Madrid for PICF collection, before any treatment is provided. This will be done with the aim of excluding potential inter-individual variability in the metabolomic and proteomic profile of PICF.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Peri-implant diseases presence | Baseline (cross-sectional part)
  Presence or absence of peri-implant mucositis or peri-implantitis according to the 2017 World Workshop (Berglundh et al. 2018)
Disease resolution of peri-implantitis | 1-year after treatment (longitudinal part)
  According to the criteria proposed by Sanz & Chapple (2012)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, University Complutense Madrid, Spain, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided